CLINICAL TRIAL: NCT04759118
Title: Effect of Prenatal Childbirth Program on Maternal Anxiety, Maternal-Fetal Attachment,
Brief Title: The Effectiveness of Modified Childbirth Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endang Koni Suryaningsih (Other)
Responsible Party: Sponsor-Investigator, Endang Koni Suryaningsih, Principal Investigator, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1303/KEP-UNISA/XI/2019
Record Dates: First submitted 2021-02-11; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Nursing Caries
Keywords: Randomized control trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The participant in his group is a pregnant woman. The facilitators of the control groups were midwives who are already providing prenatal education classes at the clinics. The classes followed the government curriculum, which consists of three classes per month and does not invite husbands to participate. However, in this study, participants in the control group have four classes over a one-month period to better match the program of the intervention group. The material for the standard curriculum includes anatomical and physiological changes during pregnancy, pregnancy care, birth, and postpartum care. The classes also address family planning after giving birth, newborn care, preventing infectious disease, and procedures for obtaining a birth certificate. The midwives also discuss and debunk unhealthy local myths, beliefs, and cultural practices surrounding pregnancy, childbirth and the postpartum period
- Experimental group (Experimental): The modified childbirth education program was applied in the experimental group. the intervention covered modification of content material, learning methods, and involving husband or other relatives during the class.
  Interventions: Behavioral: modified childbirth education program

INTERVENTIONS:
Behavioral: modified childbirth education program — The participants in the intervention group are pregnant women and their husbands. The instructors employed teaching methods such as a group discussion, watching videos, and brainstorming, as well as questions and answer periods, demonstrations, childbirth simulation, and practice. The primary investigator (PI) will teach particular sessions, including maternal-fetal attachment skills, parenting skills, comfort measures, childbirth positions, as well as knowledge about anatomy and physiology during pregnancy and birth Classes consisted of 120-minute sessions held once a week for four weeks.
  Arms: Experimental group

SUMMARY:
A randomized control trial to test the effectiveness of childbirth education programs on maternal anxiety, maternal-fetal attachment, childbirth self-efficacy, and marital satisfaction based on Roy Adaptation Model. The modified childbirth education class as the experimental group was set up by PI following health authority guidelines in Indonesia. the measurement variable outcomes in the experimental group were compared to the control group after 4 weeks of intervention. statistical analysis applied to compare demographic characteristics between two groups as well as to compare the mean score of the variable between two groups.

DETAILED DESCRIPTION:
The curriculum of the modified childbirth education (CE) program was created along with suggestions and recommendations from experts. The participants were recruited from five different health centers in Yogyakarta. the computer random block size was applied to determine the randomization (sequence 4,6,8) and allocation concealment was assured by using sequentially numbered, opaque, sealed envelopes. The participants in the intervention group are pregnant women and their husbands. The instructors employed teaching methods such as a group discussion, watching videos, and brainstorming, as well as questions and answer periods, demonstrations, childbirth simulation, and practice. The primary investigator (PI) will teach particular sessions, including maternal-fetal attachment skills, parenting skills, comfort measures, childbirth positions, as well as knowledge about anatomy and physiology during pregnancy and birth. The materials and learning methods as the control process are expected to influence the four modes as the effectors that can reduce maternal anxiety and increase maternal-fetal attachment, childbirth self-efficacy, as well as marital satisfaction as the outcomes of adaptation level. The study setting for the intervention group was conducted at the antenatal care laboratory of 'Aisyiyah University of Yogyakarta. For safety and protocol concerns during the pandemic Corona Virus Disease-19 situation, the class was set up in a big classroom and adequate ventilation that can accommodate 12 couples and is equipped with yoga mats and pillows, as well as convenient access to a restroom. The couples and researcher team were required to wear masks and wash their hand before and after entering the class. Research assistants printed handouts and lead the group through WhatsApp application to following up practicing skills at home and also respond to the question from the participant at any time. During the intervention, the health workers from the participating health centers have been invited to observe the intervention. Classes consisted of 180-minute sessions held once a week for four weeks

The control group participants in this study have attended standard childbirth education classes during the same period as the intervention group. The control group classes were conducted at the primary health centers where they were recruited, not at the university. The facilitators of the control groups were midwives who are already providing prenatal education classes at the clinics. The classes followed the government curriculum, which consists of three classes per month and does not invite husbands to participate. However, in this study, participants in the control group have four classes over a one-month period to better match the program of the intervention group. The material for the standard curriculum includes anatomical and physiological changes during pregnancy, pregnancy care, birth, and postpartum care. The classes also address family planning after giving birth, newborn care, preventing infectious disease, and procedures for obtaining a birth certificate. The midwives also discuss and debunk unhealthy local myths, beliefs, and cultural practices surrounding pregnancy, childbirth, and the postpartum period. For the fourth class, the control group has a half-hour to fill out the questionnaires and a half hour for feedback and discussion. Then the researcher and assistants have provided the control group participants with a condensed two-hour class of prenatal yoga, comfort measures, and maternal-fetal attachment activities. We conducted online briefing sessions with midwives who are the childbirth education program facilitator at five health centers. The briefing discussed the objectives of the study, the administration of the questionnaire, and the quality control issues relating to biases, fabricated data, missing data, and ethical issues. These were established in an effort to ensure consistency in the process of data collection.

ELIGIBILITY:
Inclusion Criteria:

1. First-time pregnancy (nullipara)
2. Gestational age of 28 to 35 weeks
3. Married
4. Residents of Yogyakarta
5. Singleton pregnancy

Exclusion Criteria:

* Mothers who miss the classes more than two times is considered to be excluded in the study. The mothers those who miscarry, and those whose pregnancies become high-risk, will be automatic excluded from the study

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Maternal anxiety | four weeks
  Pregnancy-related anxiety is defined as worries, concerns and fears about pregnancy, childbirth, and health of infant and future parenting. This outcome was measured using Pregnancy Related Anxiety Quistionnaire-Revised 2, developed by Van Den Bergh. consists of a 10-item self-report for multipara women, and an 11-item self-report for nulliparas. The scores on each item range from 1 (definitely not true) to 5 (definitely true). The 10-items consist of three subscales: items 1, 2, 6 and 8 are related to "fear of giving birth," items 4, 9, 10, and 11 are related to "worries about bearing a physically or mentally handicapped child," and items 3, 5, and 7 are related to body image or "concern about own appearance."The item 8 ("I am anxious about the delivery because I have never experience one before") will apply in this study since all the proposed participant are nulliparous, instead of item 1 ("I am anxious about the delivery").
Maternal-fetal attachment | Four weeks
  The unique relationship between mother and unborn baby. This relationship is progress in line the number of gestation week since the mother will experience the presence of fetal movement. This outcome is assessed using Prenatal Attachment Inventory (PAI) developed by Muller. The instrument consist of 21 Likert-type items ranging from 1 ('almost never') to 4 ('almost always'). All items are summed for a single score, and the possible range of scores is 21-84. The author have culturally translated, produce the Indonesian version of PAI, and demonstrates high internal consistency.
Childbirth Self-efficacy | Four weeks
  The maternal coping ability regarding her confidence during childbirth. This outcome was assessed using Childbirth Self-Efficacy Inventory developed by Lowe. The instrument consist of 60 items divided to four subscales; OAL, ESS, OSS and ESS. A total Childbirth Outcome Expectancy Score (Outcome-Total) is computed by summing the Outcome-AL and Outcome-SS scale scores. A Total Self-Efficacy Expectancy Score (Efficacy-Total) is computed by summing the Efficacy-AL and Efficacy-SS scale scores. The example item: " Relax my body", " tell myself that I can do it", and "listen to encouragement from the person helping me."
Marital Satisfaction | Four weeks
  The outcome of marital satisfaction was measured using Evaluation and Nurturing Relationship Issues, Communication and Happiness (ENRICH) Marital Satisfaction Scale (EMS) was developed by Fower and Olson. The tool consist of a 15-item comprising the Idealistic Distortion (5 items) and Marital Satisfaction Scales (10 items). This scale is a Likert-type ranging from 1 (strongly disagree) to 5 (strongly agree) which is consist of positive and negative statement that indicate items scored direction. Items scored in negative direction would be reverse-scored (i.e if it is mark 5, it would be scored 1; it is marked 4, it would be scored 2; a 3 remain unchanged). The EMS Scale provides a score for each partner.

CONTACTS AND LOCATIONS:
Overall Officials: Endang K Suryaningsih, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Universitas 'Aisyiyah Yogyakarta, Yogyakarta, Indonesia